CLINICAL TRIAL: NCT05413928
Title: Effect of Meal Composition and Timing Modification on Glucose Metabolism, Body Temperature and Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heyjun Park, Protocol Director, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 61843
Record Dates: First submitted 2022-05-09; First posted 2022-06-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: PreDiabetes; Type 2 Diabetes; Healthy
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will undergo a baseline phase for 20 days, where they will follow their regular dietary intake, physical activity, and sleep. They will be wearing a CGM and an activity monitor and for a couple of nights, they will use a sleep monitor. That will be followed by 4 interventional phases where they will be asked to limit their daily eating to 10 hours or less (Time Restricted Eating, TRE), with the eating window and the caloric distribution will be shifted during each of the next 3 phases, each phase lasting 20 days. The last phase will last 8 days and participants will be asked to consume provided meals with a determined amount of protein, carbohydrates, and fat. Their body temperature will be measured using a continuous temperature device and a heart rate monitor to capture dynamic rage of the sympathetic response during and after the meal consumption (thermotyping).
  Interventions: Behavioral: Time Restrictive Eating- late; Behavioral: Time Restrictive Eating- early; Behavioral: Time Restrictive Eating- early with early caloric intake; Other: Macronutrient-controlled meals

INTERVENTIONS:
Behavioral: Time Restrictive Eating- late — Eating window will be 10 hours or less, starting 3 hours after waking up. Same monitoring as Baseline phase.
Behavioral: Time Restrictive Eating- early — Eating window will be 10 hours or less, starting 30 min after waking up. Same monitoring as Baseline phase.
Behavioral: Time Restrictive Eating- early with early caloric intake — Same as TRE-early, but concentrating caloric intake early in the eating window Same monitoring as Baseline phase.
Other: Macronutrient-controlled meals — Meals with a determined amount of protein, carbohydrates, and fat.

SUMMARY:
The purpose of our study is to understand the impact of different meal timing alterations on blood sugars, metabolism, microbiome and sleep physiology in people with prediabetes and diabetes; and to study the temperature/heart rate response to different meals in different people.

DETAILED DESCRIPTION:
Pilot data points to an effect of the time between waking up and first meal is important in blood glucose management through the rest of the day. The investigators are interested in understanding the effect of caloric distribution through the day, specifically consuming more later in the day versus earlier in the day. The investigators want to test the hypothesis that consolidating the meals during a shorter span in the day (time restricted eating) can ameliorate blood sugars and sleep parameters in the studied population. The researchers would also like to compare dynamic range of meal-induced sympathetic responses (e.g. temperature and heart rate changes) between different metabolic health conditions (e.g. insulin sensitive vs insulin resistant vs diabetes) while controlling for dietary intake. Previous research studies suggest that people with different metabolic health conditions would have different meal-induced sympathetic responses. Based on this, the primary goal of the study is to characterize metabolic health based on non-invasive wearable sensor data that measure these responses.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older;
* Not be pregnant, if female;
* Be generally healthy (with no apparent symptoms at the time of enrollment)
* Patients with prediabetes or diet- controlled or type 2 diabetes or controlled with metformin, will also be allowed to participate.
* Be willing to provide written informed consent for all study procedures.

Exclusion Criteria:

* major organ disease
* pregnant/lactating
* diabetes medications except for metformin
* malabsorptive disorders like celiac sprue
* heavy alcohol use
* use of weight loss medications or specific diets
* weight change >2 Kg in the last month
* history of bariatric surgery
* Any medical condition that physicians believe would interfere with study participation or evaluation of results
* Mental incapacity and/or cognitive impairment on the part of the patient that would preclude adequate understanding of, or cooperation with, the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic control as measured by change in blood sugar values. | 5 months
  Change in glycemic control measured from baseline through all phases of study. Glycemic control is derived from continuous glucose monitor (CGM) data and expressed in milligrams/deciliter
Core body temperature response to meal consumption | Analysis of response to all standard meals will take 9 days
  Analysis of core body temperature response as measured by change from overnight fasting condition to the peak value within 4 hrs following the standardized meal consumption. Core body temperature response is derived from CTM data and expressed in Celsius.

SECONDARY OUTCOMES:
Change in sleep quality measured as duration of sleep stages | 5 months
  Duration of each sleep stage (i.e. light, deep, REM, wake stages) overnight. Sleep quality will be measured via a headband wearable device. Sleep quality will be compared to baseline through the other intervention phases.
Change in sleep quality measured as frequency of sleep stages | 5 months
  Frequency of each sleep stage (i.e. light, deep, REM, wake stages) overnight. Sleep quality will be measured via a headband wearable device. Sleep quality will be compared to baseline through the other intervention phases.
Change in wake duration during sleep | 5 months
  Measurement of Wake After Sleep Onset (WASO) in minutes. Measured via a headband wearable device. WASO will be compared to baseline through the other intervention phases.
Sleep efficiency | 5 months
  Sleep efficiency will be calculated by the following formula: 100-((WASO/total sleep duration)x100).
  Changes will be compared from baseline to the rest of the intervention phases.
Sleep latency | 5 months
  Sleep latency is the duration in minutes from being awake to falling asleep. Changes in sleep latency will be compared from baseline to the rest of the intervention phases.
Heart rate response to meal consumption | Analysis of response to all standard meals will take 9 days
  Heart rate response to meal consumption as measured by the change in heart rate from baseline (overnight fasting condition) to the peak value within 4 hrs following the standardized meal consumption. Heart rate response is derived from continuous heart rate monitoring (CHRM) data and expressed in beats per minute (bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Snyder, PhD, Principal Investigator — Stanford University; Heyjun Park, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No